CLINICAL TRIAL: NCT02456753
Title: Assesment by Ultrasonography of the Perineal-cephalic Distance in Consistence With the Notion of Clinical Fetal Head Engagement
Brief Title: Assesment by Ultrasonography of the Perineal-cephalic Distance
Acronym: ECHOTRANS
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0024
Record Dates: First submitted 2015-04-13; First posted 2015-05-28 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Ultrasonography, Prenatal
Keywords: in labor; Ultrasonography; clinical examination; Prenatal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- trans-perineal ultrasonography: Patients included are women about to give birth, they undergo a clinical examination done by midwives. Followed by a trans-perineal ultrasonography examination done by a technical operator in order to measure the perineal-cephalic distance.
  These examination are done the day of enrollment, they last for a few minutes and no further tests will be done afterwards.
  Interventions: Device: trans-perineal ultrasonography

INTERVENTIONS:
Device: trans-perineal ultrasonography — Assesment of the fetal head-perineum distance via a trans-perineal ultrasonography

SUMMARY:
The practice of ultrasounds increases in delivery rooms every year. Indeed, this method can help to visualize elements that may not be observable after clinical examination. Moreover, it is known that a fetal head engagement can lead to an instrumental extraction and in case of error, which happens in some cases, fetal and maternal risks are possible.

These elements led to the investigators' hypothesis which is that a trans-perineal ultrasonography may facilitate the evaluation of a clinical fetal head engagement in case of doubt.

DETAILED DESCRIPTION:
It's a monocentric, transversal, clinical trial regarding women giving birth at the GHICL's hospital Saint Vincent de Paul.

Clinical examinations will be done by the midwives following the indications given on the clinical form. A trans-perineal echography will then be done by technical operators following the ultrasonography form.

These examinations will only last a few minutes, no further tests will be done afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years old or older
* Primiparous
* Complete dilation of the cervix
* Gestational age of 37 weeks or more according to the date of amenorrhea - - Rupture of membranes
* Fetus in cephalic presentation
* Patient who has signed a consent form

Exclusion Criteria

* Patient for whom the fetus has died in uteri
* Patient who's coming for an abortion
* Fetus in breech or transverse presentation
* Gemellary pregnancy for which the fetus present a severe cardiac anomaly
* Patient under trusteeship or guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included are women about to give birth, they undergo a clinical examination done by midwives. Followed by a trans-perineal ultrasonography examination done by a technical operator in order to measure the perineal-cephalic distance.
  These examination are done the day of enrollment, they last for a few minutes and no further tests will be done afterwards.
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Perineal-cephalic distance measured in milimeters | one day
  Determine the perineal-cephalic distance via echographic examination, which gives a better sensitivity/specificity in comparison to the clinical examination considered as a gold standard

SECONDARY OUTCOMES:
Perineal-cephalic distance measured in milimeters according to specific conditions: posterior positions, th etime from induction to delivery, presence of caput succedaneum | one day
  Determine the interest of the echography measurement in specific conditions (variety of posterior presentations, caput succedaneum, work stagnation) regarding the diagnosis of engagement, in case of doubt concerning the clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Desurmont, MD, Principal Investigator — Groupment des Hôpitaux de l'Institut Catholique de Lille
Locations (1):
- Hôpital Saint Vincent de Paul (GHICL), Lille, Hauts-de-France, France